CLINICAL TRIAL: NCT07406373
Title: The Effect of Intra-abdominal Pressure and Abdominal Circumference on Sensory Block Level After Spinal Anesthesia in Pregnant Women Undergoing Cesarean Section
Brief Title: Intra-abdominal Pressure, Abdominal Circumference, and Spinal Block Level in Cesarean Section
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Serkan TELLİ, Assistant Professor, Kutahya Health Sciences University
Other Study IDs: 2025/08-28
Record Dates: First submitted 2026-01-23; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cesarean Section; Pregnancy; Elective Cesarean Section
Keywords: spinal block; obstetric anesthesia; sensory block level; spinal anesthesia; intra-abdominal pressure; abdominal circumference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Spinal anesthesia is commonly used for cesarean section and provides effective anesthesia with rapid onset. However, the spread of spinal anesthesia may vary among pregnant women due to physiological and anatomical changes during pregnancy. Increased intra-abdominal pressure and abdominal circumference may influence cerebrospinal fluid dynamics and affect the level of sensory block achieved after spinal anesthesia.

This prospective observational study aims to evaluate the relationship between intra-abdominal pressure, abdominal circumference, and the maximum sensory block level following spinal anesthesia in pregnant women undergoing cesarean section. Intra-abdominal pressure and abdominal circumference will be measured before surgery, and sensory block levels and hemodynamic parameters will be assessed after spinal anesthesia. The findings of this study may help to better understand factors affecting spinal block spread in pregnant patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-40 years
* Scheduled for elective cesarean section at Kütahya City Hospital
* Planned spinal anesthesia
* ASA physical status II-III
* Provided written informed consent

Exclusion Criteria:

* Refusal to participate in the study
* Emergency cesarean section
* Preeclampsia or other hypertensive disorders of pregnancy
* Onset of labor or premature rupture of membranes
* Clinical conditions affecting intra-abdominal pressure, including peripheral edema or ascites
* Height <140 cm or >180 cm
* Body mass index < 40 kg/m²
* Spinal deformity or history of spinal surgery
* Contraindications to neuraxial anesthesia
* Known allergy to bupivacaine
* Requirement for additional surgical procedures other than cesarean section
* Conditions contraindicating or interfering with intra-abdominal pressure measurement, including active or previous postdural puncture headache, neurogenic bladder, hematuria, or incidental abdominal mass

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study includes pregnant women aged 18-40 years who were scheduled for elective cesarean section under spinal anesthesia at the Department of Obstetrics and Gynecology, Kütahya City Hospital. Eligible participants belonged to ASA physical status II-III and provided informed consent. The study population represents a clinically stable obstetric cohort undergoing elective cesarean delivery, without conditions known to significantly alter intra-abdominal pressure or spinal anesthesia characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Maximum sensory block level after spinal anesthesia | Within the first 30 minutes after spinal anesthesia
  The maximum dermatomal level of sensory block assessed by loss of cold sensation after spinal anesthesia.

SECONDARY OUTCOMES:
Intra-abdominal pressure | Baseline (preoperative, before spinal anesthesia) and early postoperative period (within 30 minutes after cesarean section)
  Intra-abdominal pressure measured in the preoperative period before spinal anesthesia and in the postoperative period following cesarean section using an intravesical measurement technique.
Abdominal circumference | Baseline (preoperative, before spinal anesthesia) and early postoperative period (within 30 minutes after cesarean section)
  Abdominal circumference measured at the level of the umbilicus before spinal anesthesia and in the postoperative period following cesarean section.
Incidence of hypotension after spinal anesthesia | Within the first 30 minutes after spinal anesthesia
  Hypotension defined as mean arterial pressure <65 mmHg measured during the first 30 minutes after spinal anesthesia.
Vasopressor requirement | Perioperative period
  Requirement and total dose of vasopressor agents administered after spinal anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Şehir Hastanesi, Kütahya, Kütahya, Turkey (Türkiye)